CLINICAL TRIAL: NCT05922527
Title: Clinical and Radiographic Evaluation of Using Amnion Chorion Membrane Combined With Allograft Bone Putty for the Management of Intrabony Defects in Patients With Chronic Periodontitis: a Randomized Clinical Trial
Brief Title: Amnion Chorion Membrane Combined With Allograft Bone Putty for the Management of Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Samy Abdelmalak Hanna, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERIO2:5:1
Record Dates: First submitted 2023-06-07; First posted 2023-06-28 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Periodontal Regeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined regenerative technique (Experimental): Open flap debridement combined with Amnion Chorion Membrane and DFDBA
  Interventions: Procedure: Combined regenerative technique
- Open flap debridement (Active Comparator): Open flap debridement
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Procedure: Combined regenerative technique — Periodontal regenerative technique using amnion chorion membrane combined with DFDBA in a putty form
  Arms: Combined regenerative technique
Procedure: Open flap debridement — Open flap debridement
  Arms: Open flap debridement

SUMMARY:
The ultimate goal for periodontal management is to obtain true periodontal regeneration. Periodontal regeneration implies that CAL gain is achieved through the formation of new cementum and new inserted periodontal ligaments, accompanied by alveolar bone formation, thus a whole new periodontal apparatus is reconstructed. Combined periodontal regenerative therapy; including bone grafting are considered a viable treatment option and result in significantly better clinical outcomes in intrabony defects compared to monotherapy.

This study was conducted as a randomized controlled clinical trial to evaluate clinically and radiographically the possible predictable results regarding the use of amnion chorion allograft (ACM) barrier and demineralized freeze dried bone allograft, (DFDBA) versus open flap debridement (OFD) in treatment of periodontal intrabony defects.

DETAILED DESCRIPTION:
True periodontal regeneration is the ultimate goal for periodontal management, implies that clinical attachment level gain is achieved through the formation of new cementum and new inserted periodontal ligaments, accompanied by alveolar bone formation, thus a whole new periodontal apparatus is reconstructed. Various techniques and biomaterials have been used to achieve periodontal regeneration of intraosseous defects.

In order to compare the effectiveness of various periodontal regenerative therapies in treating periodontal infrabony defects many systematic reviews were carried out. The use of guided tissue regeneration (GTR) and the combined therapies as regenerative approaches were shown to be more effective than flap procedures, nonetheless, the differences between regenerative therapies to be minor and insignificant.

Amnion chorion placental derived membrane (ACM) has been introduced in periodontal regenerative therapy owing to its biological properties. It is biocompatible, biodegradable and promotes proliferation and migration of the adjacent autogenous connective tissue. There is no single reported incidence of graft rejection, disease transmission or immune response from using placental tissues since its first documented usage till today. ACM has been used in many surgical dental procedures as GTR, alveolar bone preservation and guided bone regeneration. ACM possesses unique features that make it different from other materials used in this fields. In periodontal regenerative procedures as GTR, ACM assists rapid epithelial cell growth instead of epithelial cells exclusion as for the traditional concept of GTR. As epithelial cells are encouraged to migrate rapidly across the ACM barrier, they form an epithelial seal over the underlying bone graft or bony defect space and do not apically migrate into the defect .

Several studies support the use of ACM as an effective material alternative to the currently used materials/techniques for periodontal regeneration procedures, however more well conducted studies are still needed.

Accordingly, numerous data and researches are available nowadays, which support the great and variant regenerative capacities of the different periodontal biomaterials that are widely available and currently used for treatment of periodontal intra-bony defects, especially DFDBA and ACM. However, minimal radiographic findings were mentioned in the previous systematic reviews comparing combined regenerative approach and OFD.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent tooth.
* Tooth with two or three-walled intra-bony defect, PPD ≥ 5mm with intra osseous defect ≥ 3mm.
* Good oral hygiene.
* Compliance with the maintenance program.
* Accepted the 6 months follow-up period.

Exclusion Criteria:

* Teeth with one wall intra-bony defect or supra-bony defects.
* Teeth with grade II or III mobility.
* Teeth with proximal carious defects or proximal faulty restorations.
* Medically compromised patients.
* Pregnant or nursing women.
* Smokers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level gain | 6 months
  clinical attachment level gain intragroup and intergroup, measured clinically in mm using periodontal probe

SECONDARY OUTCOMES:
Probing Pocket Depth Change | 6 months
  Probing pocket depth change, measured clinically in mm using periodontal probe
Bone defect area | 6 months
  bone defect area, measured radiographically in mm3 using periapical radiographs

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt